CLINICAL TRIAL: NCT01842971
Title: Associating Liver Partition and Portal Vein Ligation (ALPPS) for Potentially Resectable Liver Metastasis From Colorectal Cancer: Prospective Evaluation of the Early Two-stage Hepatectomy by the Simon's Methods
Brief Title: ALPPS (Liver Partition and Portal Vein Ligation) for Two-stage Hepatectomy for Colorectal Liver Metastasis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Main reason: negative echo in the literature after the first publications.
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2012_843_0028; A41707-36 (Other: french ANSM)
Record Dates: First submitted 2013-04-24; First posted 2013-04-30 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
Keywords: two stage hepatectomy; liver metastasis; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- two stage hepatectomy (Experimental): the two stage hepatectomy is defined as a two step procedure: first step: hepatotomy with ligature of the right branch of the portal vein second step (one week after the first step): right hepatectomy
  Interventions: Procedure: two stage hepatectomy

INTERVENTIONS:
Procedure: two stage hepatectomy

SUMMARY:
The aim of this study is evaluate the feasibility of early two-stage hepatectomy in patients with liver metastasis from colorectal cancer.

DETAILED DESCRIPTION:
In France, each year around 36,000 new cases of colorectal cancers are registered responsible in 16,000 deaths because of liver metastasis.

In case of bilobar metastasis, classic two-stage hepatectomy with portal embolization could be performed.

An alternative to the classic surgery, early two stage hepatectomy, could be proposed to simplify the patient's management and to improve the resectability.

ELIGIBILITY:
Inclusion Criteria:

* potentially resectable liver metastasis from colorectal cancer
* portal embolisation required
* older than 18 years old

Exclusion Criteria:

* synchronous surgery on the colon or the rectum
* extra hepatic metastasis
* history of hepatectomy
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
number of complete surgical procedure | postoperative week 4
  the number of complete surgical procedure is defined as the number of patients in whom the two stage hepatectomy is complete.

SECONDARY OUTCOMES:
overall mortality | one year after the two stage hepatectomy
  the overall mortality is defined as the number of patients who are dead at one year after the surgery
number of patient with hepatocellular insufficiency | postoperative day 30
  the hepatocellular insufficiency is defined by a prothrombin rate below 50%
overall morbidity | postoperative day 30
  the overall morbidity is classified according to the Dindo Clavien classification
preoperative liver volumetry | one week prior to the surgery
  the remnant liver volume is evaluated with the Myrian Software and calculated by the radiologist
quality of life | the day before the first stage surgery and the day before the second stage surgery
  the quality of life is evaluated thanks to the EORTC QLQ C30 LMC 21 form the day before the first stage surgery and the day before the second stage surgery.

CONTACTS AND LOCATIONS:
Overall Officials: jean marc regimbeau, MD, PhD, Principal Investigator — Amiens University Hospital
Locations (1):
- Amiens University Hospital, Amiens, France